CLINICAL TRIAL: NCT04218968
Title: The Effect of Adrenergic Blocker Therapy on Cardiac and Striatal Transporter Uptake in Pre-Motor and Symptomatic Parkinson's Disease: a Follow Up Study
Brief Title: Cardiac Changes in Early Parkinson's Disease: a Follow Up Study
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Michele Tagliati, MD, Professor and Vice Chairman, Director of Movement Disorders, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study00000349
Record Dates: First submitted 2019-12-26; First posted 2020-01-06 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: REM Sleep Behavior Disorder; Pre-motor Parkinson Disease; Symptomatic Parkinson Disease
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease, Secondary | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- carvedilol therapy (Experimental): Twice daily oral doses of adrenergic blocker 12.5 mg or 25mg, according to patient tolerability.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Primary procedures in this study are MIBG scan, DAT scan, NM-MRI, and carvedilol titration. Subjects will return for research visits and imaging every six months for three years. The investigators hypothesize that the rate of decline in DAT scan123I-Ioflupane uptake will be slower in subjects who have received the adrenergic blocker carvedilol, resulting in a decreased clinical phenoconversion rate to parkinsonism.

SUMMARY:
The purpose of this study is to investigate the long-term effects of treatment with the adrenergic blocker carvedilol on serial DaTscan, a dopamine transporter (DAT) single photon emission computerized tomography (SPECT) imaging technique in a population of subjects with defined pre-motor Parkinson's disease risks (i.e., REM sleep Behavior Disorder (RBD) and at least one among hyposmia, constipation, depression and color vision abnormality) and abnormal 123I-Metaiodobenzylguanidine (MIBG) scintigraphy.

DETAILED DESCRIPTION:
Primary procedures in this study are MIBG scan, DAT scan, Neuromelanin Magnetic Resonance Imaging (NM-MRI), and carvedilol treatment. Subjects will return for research visits and imaging tests every six months for three years. We hypothesize that the rate of decline in DAT scan123I-Ioflupane uptake will be slower in subjects who have received the adrenergic blocker carvedilol, resulting in a decreased clinical phenoconversion rate to parkinsonism. If this is true, it might create a considerable window of opportunity for treatment with adrenergic blockers - or similar compounds able to reduce Sympathetic Nervous System (SNS) hyperactivity - which may result in long-term benefits such as delaying the neurodegenerative process and the onset of neurological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the study "The Effect of Adrenergic Blocker Therapy on Cardiac and Striatal Transporter Uptake in Pre-Motor and Symptomatic Parkinson's Disease" (Pro#00053136)
* Capacity to give informed consent

Exclusion Criteria:

* Secondary Parkinsonism, including tardive
* Concurrent dementia defined by a score lower than 22 on the MoCA
* Concurrent severe depression defined by a BDI fast screen score greater than 13
* Comorbidities related to SNS hyperactivity

  * Heart failure (LVEF <45%)
  * Recent myocardial revascularization (<12 weeks)
  * Hypertension (SBP>150mmHg or DBP>100mmHg)
  * Chronic Atrial fibrillation
  * Concurrent Use of Beta-adrenergic antagonist
  * Diabetes mellitus
  * COPD
  * Untreated Sever Sleep Apnea; Apnea-Hypopnea Index (AHI) > 30/h.
  * Severely reduced kidney function (Glomerular Filtration Rate<30ml/min)
* Contraindications to the use of carvedilol

  * Asthma or bronchospasm
  * Recent myocardial infarction (<48 h)
  * Ongoing unstable angina
  * Cardiogenic shock or prolonged hypotension
  * Second or Third-Degree AV block
  * Significant valvular aortic stenosis
  * Obstructive cardiomyopathy, or constrictive pericarditis
  * Resting Heart Rate (RHR)< 45 Or Bradycardia (HR<60) with at least one of the following symptoms; Lightheadedness, dizziness, weakness, Altered mental status, Shortness of breath, Pre-Syncope, Syncope, Sick Sinus Syndrome, Stroke within the past 1 month, Severe Hepatic Dysfunction
* Allergy/hypersensitivity to iodine or study medication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in 123I-Ioflupane uptake - DATscan | Every year for three years
  Changes in 123I-Ioflupane uptake, as measured by specific binding ratio (SBR), between baseline, year one, year two and year three.

SECONDARY OUTCOMES:
Diagnosis of PD or other synucleinopathies by the end of 3 years in the study population | Every year for 3 years
  Clinical evaluation
Changes in 123I-MIBG late H/M | Every 6 months for 3 years
  Changes in 123I-MIBG reuptake, as measured by late H/M ratio, between baseline and every six months for three years
Changes in 123I-MIBG WR rate | Every 6 months for 3 years
  Changes in 123I-MIBG WR reuptake, as measured by WR rate, between baseline and every six months for three years
Sensitivity and specificity of DAT Scan compared to MIBG in predicting RBD conversion to PD/other synucleinopathies | Every year for3 years
  Changes in 123I-Ioflupane uptake, as measured by specific binding ratio (SBR), between baseline, year one, year two and year three.

OTHER OUTCOMES:
MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III | Every 6 months for 3 years
  MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III changes from OFF medication between baseline and every 6 months for three years
Non-Motor Symptoms Scale (NMSS) changes | Every 6 months for 3 years
  Non-Motor Symptoms Scale (NMSS) changes between baseline and every 6 months for three years
Scales for Outcomes in Parkinson's Disease - Autonomic Dysfunction (SCOPA-AUT) | Every 6 months for 3 years
  Scales for Outcomes in Parkinson's Disease - Autonomic Dysfunction (SCOPA-AUT) changes between baseline and every 6 months for three years
REM sleep Behavior Disorder Screening questionnaire (RBDSQ) | Every 6 months for 3 years
  REM sleep Behavior Disorder Screening questionnaire (RBDSQ) changes between baseline and every 6 months for three years
University of Pennsylvania Smell Identification Test (UPSIT) | Every 6 months for 3 years
  University of Pennsylvania Smell Identification Test (UPSIT) changes between baseline and every 6 months for three years
Functional constipation score changes | Every 6 months for 3 years
  Functional constipation score changes between baseline and every 6 months for three years. The total score has a range of 0 to 12, with scores > 4 identifying functional constipation
Color vision changes | Every 6 months for 3 years
  Color vision changes, as assessed using HRR Pseudoisochromatic Plates, between baseline and every 6 months for three years
Central and peripheral insulin resistance changes | Every 6 months for 3 years
  Peripheral Insulin Resistance (IR) will be defined by testing for fasting plasma insulin (FPI), fasting plasma glucose (FPG) and glycated hemoglobin (HbA1c). HOMA index will be calculated by the formula: HOMA-IR = (FPI x FPG)/405 . A cutoff HOMA index of 2.0, equivalent to <50% sensitivity, will be used to define IR. Subjects were considered to have IR if they either had a HOMA≥2.0 and/or HbA1c≥5.7 . In addition, measures of insulin sensitivity in neuronal-origin enriched plasma EVs (central IR) will be used to test the association of changes in such sensitivity to changes in MIBG uptake and clinical scores from baseline and every 6 months. For that purpose, plasma samples will be collected and stored and -80oC to allow for isolation of neuronal origin EVs at the completion of the study
Differences in integrity of pigmented neurons in the locus coeruleus and substantia nigra between baseline, year one, year two and year three | 3 years
  This outcome will be measured by the content of neuromelanin, a product of cathecolamine metabolism in LC and SN.
Correlation between changes in integrity of pigmented neurons of substantia nigra as measured by neuromelanin-sensitive magnetic resonance imaging (MRI) and 123I-Ioflupane uptake as measured by Dopamine Transporter Imaging (DAT scan) | 3 years
  These measurements will be aggregated to calculate the correlation between changes in neuromelanin content as measured by NM-MRI and dopamine content as measured by DAT scan
Heart Rate Variability (HRV) changes between baseline and every 6 months for three years | Every 6 months for 3 years
  Beat-to-beat intervals will be registered to assess sympatho-vagal balance every 6 months for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michele L Lima Gregorio, MD, FAAN, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Michele L Lima Gregorio, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No